CLINICAL TRIAL: NCT01947634
Title: Cross-sectional Study on the Incidence of Sleepiness and Sleep-disordered Breathing in Patients With Fabry Disease
Brief Title: Sleepiness and Sleep-disordered Breathing in Fabry Disease. A Prospective Cohort Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SleepFabry
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ResMed Apnea Link plus (Experimental): Overnight respiratory polygraphy is performed in Fabry patients
  Interventions: Other: ResMed Apnea Link plus

INTERVENTIONS:
Other: ResMed Apnea Link plus — Overnight respiratory polygraphy to detect sleep-related breathing disorders is performed in Fabry patients

SUMMARY:
Prospective, observational cohort study to investigate the prevalence of sleepiness and sleep-related breathing disorders in patients with Fabry disease (FD). For this, an Epworth Sleepiness Score (ESS) and ambulatory overnight respiratory polygraphy (oRP) is obtained in all subjects.

DETAILED DESCRIPTION:
There are 76 patients with Fabry disease in the region of eastern Switzerland who are observed and treated in the University Hospital Zurich. All patients are encountered in retrospective cohort study, and all patients are asked to participate in the study by obtaining written informed consent.

Eligible Fabry patients are investigated by completion of ESS and one ambulatory overnight respiratory polygraphy (oRP). An ESS over 11 is defined as excessive daytime sleepiness(EDS). An apnoea/hypopnoea index (AHI) over 5 per minute is defined as sleep apnoea. Distinction of obstructive sleep apnoea (OSA) and central sleep apnoea (CSA) is performed by analysis of oRP. Medical history, clinical and laboratory data, and current treatment will be extracted from patient files and the retrospective cohort study, respectively.

The patients are asked to participate in the study at clinically regular follow-up visits. After obtaining informed consent, the subjects are provided for reviewing in- and exclusion criteria. For this, additional laboratory analyses and completion of ESS and patient's health questionnaire (PHQ-9) is required.

The screening visit is encountered in the routine clinical follow-up examination. After obtaining informed consent, the subjects are provided for reviewing in- and exclusion criteria. For this, the laboratory results (s. exclusion criteria), which are part of the routine follow-up examination, are checked, and PHQ-9 and ESS are completed together with the patient.

In case of fulfilling all inclusion criteria without presence of exclusion criteria, the patients are scheduled by telephone call for visit 1 (oRP).

Eligible Fabry patients are investigated one ambulatory overnight respiratory polygraphy (oRP). For this reason, the subjects are asked to pick-up and learn the self-administration of the oRP device (ApneaLink™ Plus (ResMed)). The oRP itself is easily performed at subject's home. The following day, the patients need to return the device, or, alternatively, they can send it by post. After oRP, there is no need for further visits for purpose of the study. The subjects are informed about the results of oRP during the next regular clinical follow-up visit.

ORP is a non-invasive medical examination technique, which is routinely applied to detect sleep-related breathing disorders. For purpose of the oRP, the ApneaLink™ Plus (ResMed), a home sleep testing diagnostic device that provides simple, cost-effective and reliable results, is applied. The subjects will be instructed in the usage of the device, so that they can install themselves in the study night.

ELIGIBILITY:
Inclusion criteria: Established diagnosis of Fabry disease, who

* are 18 years or above
* have signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Prevalence and type of sleep-related breathing disorder in Fabry patients. | Day 1
  Prevalence and type of sleep-related breathing disorder in Fabry patients measured with overnight ambulatory respiratory polygraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — University Hospital Zurich, Division of Internal Medicine
Locations (1):
- University Hospital Zurich, Division of Internal Medicine, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Franzen D, Gerard N, Bratton DJ, Wons A, Gaisl T, Sievi NA, Clarenbach CF, Kohler M, Krayenbuhl PA. Prevalence and Risk Factors of Sleep Disordered Breathing in Fabry disease: A Prospective Cohort Study. Medicine (Baltimore). 2015 Dec;94(52):e2413. doi: 10.1097/MD.0000000000002413. PMID 26717401